CLINICAL TRIAL: NCT03908112
Title: Interventions for Convergence Insufficiency in Concussed Children (ICONICC)
Brief Title: Interventions for Convergence Insufficiency in Concussed Children
Acronym: ICONICC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mitchell Scheiman (Other)
Collaborators: Ohio State University (Other); University of Alabama at Birmingham (Other); Marshall B. Ketchum University (Unknown); Stanford University (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other); New Jersey Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Mitchell Scheiman, Dean of Research, Salus University
Organization: Salus University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Salus 1003-2019
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Concussion; Convergence Insufficiency
Keywords: convergence insufficiency; concussion; vision therapy; vision rehabilitation
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: To compare the effectiveness of SC, SC+, SC plus office-based vergence/accommodative therapy for improving a composite outcome measure of clinical findings (near point of convergence and positive fusional vergence at near) in children 11-17 years of age with concussion-related CI after 12 weeks of treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be masked to the treatment assignment and at follow-up examinations the examiners will be masked to the treatment group assignment. Investigators providing the therapy will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Community Concussion Care (SC) (Active Comparator): Standard concussion care consists of physical and cognitive rest immediately following the injury for a brief period of time to allow symptoms to abate, followed by a gradual reintroduction of academic and physical activities, restricting activities at high risk for repeat brain injury (such as contact or collision sports) until a graded return to play protocol has been completed in a symptom-free manner.
  Interventions: Behavioral: Standard Community Concussion Care (SC)
- SC plus Simple Convergence Procedures (SC+) (Experimental): In addition to the treatment described for SC, participants in this group will be asked to work with the Brock String, which is a popular and simple therapy technique designed to improve convergence. A 3-phase, graded Brock String procedure has been developed for ICONICC.
  Interventions: Behavioral: SC plus Simple Convergence Exercises (SC+)
- SC plus Office-based Vergence/Accommodative Therapy (SC+VAT) (Experimental): Office-based vergence accommodative therapy (OBVAT) is administered by a study certified therapist at weekly intervals (60-minute office visits with 55 minutes of therapy time), combined with procedures to practice at home for 15 minutes, 5 times per week.
  Interventions: Behavioral: SC plus Office-based Vergence/Accommodative Therapy (SC+OBVAT)

INTERVENTIONS:
Behavioral: Standard Community Concussion Care (SC) — temporary rest, gradual increase in activity, and return to school and sports. In some cases vestibular an balance therapy are necessary, aerobic exercises, medication, counseling.
  Other Names: Concussion treatment
  Arms: Standard Community Concussion Care (SC)
Behavioral: SC plus Simple Convergence Exercises (SC+) — In addition to standard community care in this intervention the participants must perform convergence therapy every day at home
  Other Names: Concussion care plus convergence exercises
  Arms: SC plus Simple Convergence Procedures (SC+)
Behavioral: SC plus Office-based Vergence/Accommodative Therapy (SC+OBVAT) — In addition to standard community care in this intervention the participants must come to the office once a week for a 1-hour therapy session with a therapist. Office-based vergence/accommodative therapy is performed for 12 weeks with home reinforcement.
  Other Names: vision therapy
  Arms: SC plus Office-based Vergence/Accommodative Therapy (SC+VAT)

SUMMARY:
The ICONICC Study is a randomized controlled clinical trial designed to compare the proportion of successful treatment outcomes between children assigned to standard concussion care only, standard concussion care plus simple convergence procedures, or standard concussion care plus office-based vergence/accommodative therapy in children aged 11 to 17 years with symptomatic post-concussion syndrome. Children with post-concussion syndrome (4-12 weeks post-concussion injury) and symptomatic CI will be randomized to a 12-week treatment program of either standard concussion care (SC), SC plus simple convergence procedures (SC+), or SC plus office-based vergence/accommodative therapy SC+OBVAT (1:1:1 ratio).

The study will also compare the effect of treatment on clinical measures of both accommodation and vergence, symptom level/burden, health-related quality of life, clinical measures of saccadic eye movement, and objective eye movement measurements of disparity vergence, saccadic function, and accommodative function. The attainment of objective eye movement measures provides an opportunity to understand the underlying neurophysiology of the vergence and accommodative systems. Objective eye movement recordings are powerful because of the rich foundation from primate single-cell recordings that show a direct correlation with vergence and accommodative parameters in the supraoculomotor area of midbrain2, 3 and the oculomotor vermis of the cerebellum.4, 5 Thus, a combined approach of acquiring both clinical vision function measures and objective eye movement recordings in children with PCS-CI may lead to better characterization of the oculomotor phenotype with subsequent improved and personalized therapeutic interventions.

DETAILED DESCRIPTION:
Objectives:

A group of 264 diverse children, ages 11 to 17 years, with post-concussion syndrome (4-12 weeks post-concussion injury) and symptomatic CI will be enrolled from 6 sites from across the United States, will be randomized to 12 weeks of: 1) standard care (SC), 2) SC plus simple convergence exercises (SC+), and 3) SC plus office-based vergence/ accommodative therapy (SC+OBVAT).

Primary Objective: To compare the effectiveness of SC, SC+, SC plus office-based vergence/accommodative therapy for improving a composite outcome measure of clinical findings (near point of convergence and positive fusional vergence at near) in children 11-17 years of age with concussion-related CI after 12 weeks of treatment.

* Secondary outcome measures
* Objective measures of disparity vergence, accommodation, saccades, and smooth pursuit
* Quality of life measures
* Convergence Insufficiency Symptom Survey Concussion Version (CISS-CON)
* PedsQL Version 4 For participants in any treatment group who not "successful" based on the composite score described above, additional/different treatment will be offered as an option after the primary outcome examination

ELIGIBILITY:
Inclusion Criteria:

ICONICC will enroll children of all races and will adhere to a policy of equitability. To be eligible to participate in ICONICC, the child must meet all of the following criteria:

1. Medical diagnosis of concussion of at least 4 weeks and no longer than 12 weeks since known date of injury
2. Age 11 to 17 years
3. Gender - any
4. CI Symptom Survey (CISS) score ≥ 16
5. Exophoria at near at least 4∆ greater than at far
6. Receded near point of convergence (NPC) of greater than 6 cm break
7. Insufficient positive fusional vergence (PFV) at near (i.e., failing Sheard's criterion1 or PFV ≤15∆ base-out break)
8. Best-corrected distance visual acuity of 20/25 or better in each eye
9. Random dot stereopsis appreciation of 500 seconds of arc or better using the Randot Stereotest
10. Willing to wear refractive correction for any of the following uncorrected refractive errors based on a cycloplegic refraction performed at the eligibility examination. (Correction must be worn for at least 2 weeks):

    * Myopia > -0.75 D spherical equivalent in either eye
    * Hyperopia > 2.00 D spherical equivalent in either eye
    * Anisometropia > 0.75D spherical equivalent or ≥ 1.50 D in any meridian
    * Astigmatism > 1.00 D in either eye
11. Willing to discontinue BI prism or a plus add at near for duration of study (must discontinue at least 2 weeks before eligibility examination)
12. Parent and child understand protocol and are willing to accept randomization
13. Normal pupillary responses

Exclusion Criteria:

1. Any strabismus at distance
2. Constant strabismus at near
3. Limitation on versions/ductions due to restrictive or paretic strabismus
4. Esophoria of ≥ 2∆ at distance
5. Vertical heterophoria ≥ 2∆ at distance or near
6. ≥ 2 line interocular difference in best-corrected visual acuity
7. Manifest or latent nystagmus
8. History of surgery or botulinum toxin for strabismus or any type of refractive surgery
9. Previous diagnosis of CI by an eye care professional before concussion
10. Diseases known to affect accommodation, vergence, or ocular motility such as multiple sclerosis, Graves orbitopathy, myasthenia gravis, diabetes mellitus, Parkinson's disease
11. Inability to comprehend and/or perform any study-related, clinical vision function test
12. Household member enrolled in present ICONICC study or treated within the past 6 months with any form of office-based vergence/accommodative therapy or home-based vergence therapy (e.g., computerized vergence therapy)
13. Household member is an eye care professional, ophthalmic technician, ophthalmology or optometry resident or fellow, or optometry student

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Measure of the Near Point of Convergence (NPC) and Positive Fusional Vergence at Near (PFV) | 12 weeks
  To evaluate successful treatment of CI, we will use a composite outcome classification of the 2 clinical outcome measures of NPC and PFV from baseline to the primary outcome examination. A participant will be defined as successfully treated if both criteria are met: 1) normal NPC (i.e., less than 6 cm) and 2) normal PFV (i.e., greater than 15 prism diopters base-out and passing Sheard's criterion

SECONDARY OUTCOMES:
Peak velocity for 4° symmetrical convergence steps | 12 weeks
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Peak velocity will be measured with this instrument and a secondary outcome measures will be the change in peak velocity for 4° symmetrical convergence steps
Time to peak velocity for 4° symmetrical convergence steps | 12 Weeks
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in time to peak velocity for 4° symmetrical convergence steps
Latency for 4° symmetrical convergence steps | 12 weeks
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in latency for 4° symmetrical convergence steps
Response Amplitude for 4° symmetrical convergence steps | 12 weeks
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in response amplitude for 4° symmetrical convergence steps
Convergence Insufficiency Symptom Survey - Concussion Version (CISS-CON) | 12 weeks
  The change in the score on this survey will be a secondary outcome assessing symptoms
Post-concussion Symptom Inventory (PCSI) | 12 weeks
  PCSI is a 26-item validated symptom inventory for children with concussion that identifies physical, cognitive, emotional and sleep factors following injury and is useful in capturing and tracking post-injury symptoms through recovery. The change in this score will be used as a secondary outcome measure.
PedsQL (Pediatric Quality of Life Inventory) | 12 Weeks
  PedsQL (Pediatric Quality of Life Inventory) measures health-related quality of life (HRQOL) in children and adolescents. The change in this score will be used as a secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, PhD, Study Chair — Salus University
Locations (8):
- United States (8):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Marshall B. Ketchum University, Southern CA College of Optomwtry, Fullerton, California
  - Stanford University Medical Center, Palo Alto, California
  - Boston's Children's Hospital, Boston, Massachusetts
  - New Jersey Institute of Technology, Newark, New Jersey
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Salus University/Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
A number assigned centrally by the CC will identify all enrolled participants. Participant data will be secured, all clinical sites, the CC, and the Resource Center in a manner to protect participant confidentiality. Only the PI, Clinic Coordinator, and Therapist will have access to the data at the clinical site. Data will be transmitted to the CC via a secure website, with the participant identified by his/her study ID number only. The informed consent document will inform all participants that their data will be sent to the Coordinating Center. Although results of the study will be presented at scientific meetings and reported in medical journals, at no time will any of the study participants be identified. The study will be monitored by the DSMC (see below) to ensure the safety of participants.